CLINICAL TRIAL: NCT01990170
Title: Long-term Healing and Recurrence of Chronic Venous Ulcerations Following Ultrasound-guided Foam Sclerotherapy
Brief Title: Longterm Outcomes of Venous Ulcers After Foam Sclerotherapy
Status: Completed | Type: Observational
Sponsor: Heart of England NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 2013080VS
Record Dates: First submitted 2013-10-30; First posted 2013-11-21 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Chronic Venous Hypertension With Ulcer and Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ultrasound-guided foam sclerotherapy: This project is ongoing from an original study conducted by our research group looking at short- and mid-term clinical outcomes after UGFS. The original patient cohort from the aforementioned study was made up of 132 patients who underwent UGFS between 1 March 2005 and 31 December 2009 for treatment of a chronic venous ulcer (CEAP classification C5 or C6 disease) with significant (>0.5s) SVR confirmed with duplex ultrasound.

SUMMARY:
The purpose of this study is to determine long term healing rates of chronic venous ulcers (CVU) after ultrasound-guided foam sclerotherapy (UGFS) of superficial venous reflux (SVR) and to relate recurrence of CVU to evidence of recanalisation and the presence of superficial or deep venous reflux

DETAILED DESCRIPTION:
This study is attempting to follow up the original cohort of patients who took part in the short- and mid-term study which may mean reduced patient numbers due to some inevitable patient deaths. Kaplan-Meier analysis will control for this. In terms of patient numbers, effort will be made to recruit as many patients as possible as this will increase the validity of the results. This could be a problem not only related to deaths of some of the patients but also the timeframe for completion of the project or a refusal of the patient to take part. Many of the patients are elderly and may not want to accept the invitation to come to the hospital. However, good follow-up rates were achieved in the mid-term study (around 80%) and familiarity with the team should aid recruitment as the same patients will be contacted.

In order to maintain validity and reliability of the study as part of a follow on, the methodology adopted for this project will be similar to that of the short-term study in terms of the way in which the information is gathered and the classification of the results. This will mean that if a comparison between the two is to be made, similar information is available and scientifically comparable. There should not be any significant intra and/or inter observer/operator variability with the results (different users technical ability with ultrasound) as collaboration between those responsible for collection of all the data and performing all diagnostic tests will be done to avoid any potential problems with validity. For this reason, assessments will be performed by the principal investigator under the guidance and supervision of the main research nurse responsible for data collection on the previous project. Results of this study will be analysed, evaluated and disseminated as a continuation of the previous short/mid-term study.

A possible limitation may be that patient recollection of their experience of any ulcer recurrences may be unreliable. This is an unavoidable problem but effort will be made to get the most accurate account as possible from the participants.

There is a possibility for bias of the long-term follow up results as it is more likely that patients who are having problems with their treatment results will accept the offer of additional follow-up rather than those patients who are fine. However, as all patients will be asked if they would like to participate via telephone if unwilling to come to the hospital for assessment, this should not affect research question 1.

ELIGIBILITY:
Inclusion Criteria:

All patients who are unwilling or unable to consent will be excluded from the project. Any patients who have died since the mid-term study will not be contacted. All patients who are willing to attend will be entered into both outcome arms of the study analysis (see endpoints at the end of this section) and those who are unable to attend for an appointment but wish to take part will be posted a consent form and then entered into endpoint analysis 1.

-

Exclusion Criteria:

N/A

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at Heart of England NHS Foundation Trust who took part in a previous study investigating Chronic Venous Ulcers.
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2013-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Ulcer-free survival following UGFS for the treatment of CVU | Up to 5 months

SECONDARY OUTCOMES:
Superficial/deep venus reflux-free survival following UGFS for CVU | up to 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Katy Bloom, MRes, Principal Investigator — Heart of England NHS Trust
Locations (1):
- Heart of England NHS Foundation Trust, Birmingham, West Midlands, United Kingdom